CLINICAL TRIAL: NCT06087757
Title: Clemastine Treatment in Individuals With Williams Syndrome- a Double-blind Placebo Control to Assess the Safety and Efficacy
Brief Title: Clemastine Treatment in Individuals With Williams Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Prof. Doron Gothelf MD, Head of The Child and Adolescent Psychiatry Unit, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 9011-21-SMC
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Williams Syndrome
Keywords: Clemastine; Cognition; Myelination abnormalities
MeSH Terms: conditions — Williams Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is an open-label study with a blinded randomized withdrawal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Label (Experimental)
  Interventions: Drug: Open Label Clemastine with a blinded randomize withdrawal
- Blinded randomize withdrawal (Experimental)
  Interventions: Drug: Open Label Clemastine with a blinded randomize withdrawal

INTERVENTIONS:
Drug: Open Label Clemastine with a blinded randomize withdrawal — Clemastine will be given in doses as the maximum dose recommended for allergy condition. Age 6-12 years 4.02 mg/day, age 12-30 years 8.04 mg/day.

SUMMARY:
This study explores the neurobiological etiology of Williams syndrome and potential therapeutic targets for associated social, motor, and cognitive abnormalities. The main translational objective will be to test the effectiveness of Clemasntine on neurocognitive and other associated abnormalities in individuals with Williams syndrome.

DETAILED DESCRIPTION:
The overarching aim of the research proposed is to examine the safty of Clemastine use for individuals with Williams syndrome. Further, we wish to examine the relationship between Clemastine treatment and cognitive, motor and behavioral deficits in individuals with Williams syndrome. This study is an open-label study with a blinded randomize withdrawal. Each participant will go through a baseline evaluation (see study outcomes) and will be treated with the FDA approved drug Clemastine, in an age dependent dose (dosage table below). After a substantial improvement will be noticed, the participants will be divided into 2 groups, in a randomized, double-blind, placebo-control study design.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Williams syndrome, which has been confirmed by genetic testing.
* Ages 6-30.
* Normal values in safety variables (e.g. Normal ECG 120-129/80-84).
* No change in psychotropic medications and dosage during the last 4 weeks.
* During the study, no pharmacological change that may impact the study (e.g. ADHD
* medications).

Exclusion Criteria:

* Individuals with another genetic disorder besides Williams syndrome.
* Individuals with Williams syndrome, younger than 6 or older than 30 years old.
* Significant change in normal values in safety variables (e.g. high or low ECG).
* Change in medications and dosage during the last 4 weeks prior the beginning and
* during the study.
* Pregnancy.
* Using addictive substances such as alcohol.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive measures | December 2024
  Wechsler Intelligence Scale: The standard age-appropriate Wechsler scale. Wechsler Intelligence Scale for Children, 4th edition(Wechsler 1991, Wechsler 2003) for subjects 17 years and younger and the Wechsler Adult Intelligence Scale, 3rd edition (WAIS III)(Wechsler 1997) for subjects older than 17 years.
  NIH ToolBox (NIHTB): the NIHTB is a computerized neurocognitive battery developed by NIH that was designed to include measures of cognitive flexibility and inhibitory control, as well as a measure of working memory. http://www.healthmeasures.net/explore-measurement-systems/nih-toolbox/

SECONDARY OUTCOMES:
Motor and Neurological assessment. Motor and Neurological assessment. Motor and Neurological assessment. Motor and neurolocgial measures | December 2024
  The Beery-Buktenica Developmental Test of Visual-Motor Integration
  GAITRite walkway: GAITRite is a sensitive walkway measuring temporal and spatial parameters.
  Psychiatric evaluation: a semi-structured interview for neuropsychiatric diagnoses with the Schedule for Affective Disorders and Schizophrenia for School-Aged Children.
  The Child Behavior Checklist: measures behavioral/emotional problems and competencies.
  Attention Deficit Hyperactivity Disorder Rating Scale.
  The Screen for Child Anxiety-Related Emotional Disorders.
  The Social Responsiveness Scale-Second Edition.
  Adaptive Behavior Assessment System-2nd Edition.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Child and Adolescent Psychiatry Unit, Sheba Medical Center, Ramat Gan
  - Tel Aviv University, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided